CLINICAL TRIAL: NCT03368092
Title: A Prospective, Randomized Multicenter, Double Blind Clinical Trial Comparing Inhaled Dornase Alfa and Its Placebo to Reduce the Incidence of Moderate to Severe ARDS in Ventilated Trauma Patients in the Intensive Care Unit
Brief Title: Inhaled Dornase Alpha to Reduce Respiratory Failure After Severe Trauma
Acronym: TRAUMADORNASE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6998
Record Dates: First submitted 2017-12-04; First posted 2017-12-11 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Multiple Trauma; Respiratory Distress Syndrome, Adult
Keywords: severe trauma; acute respiratory distress syndrome; damage-associated molecular patterns; neutrophil extracellular traps; dornase alfa
MeSH Terms: conditions — Multiple Trauma; Respiratory Distress Syndrome; Wounds and Injuries | interventions — dornase alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dornase alfa (Experimental): Dornase alfa (Pulmozyme®, Roche 2500U, 2,5mL) given by aerosol in the respiratory circuit (Aerogen solo®) within 6h at day 1 and 24 hours after on day 2.
  Interventions: Drug: Dornase Alfa Inhalant Solution [Pulmozyme]
- Placebo (Placebo Comparator): NaCl 0,9%, given by aerosol in the respiratory circuit within 6h at day 1 and 24 hours after on day 2.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Dornase Alfa Inhalant Solution [Pulmozyme] — Dornase alfa (Pulmozyme®, Roche 2500U, 2,5mL) given by aerosol in the respiratory circuit (Aerogen solo®) within 6h at day 1 and 24 hours after on day 2.
  Arms: Dornase alfa
Drug: Placebos — NaCl 0,9%, given by aerosol in the respiratory circuit within 6h at day 1 and 24 hours after on day 2.
  Arms: Placebo

SUMMARY:
Severe hypoxemia following trauma may happen in many circumstances (aspiration, ventilation-associated pneumonia, lung contusion...), most of which are not exclusively associated with a direct injury to the lungs. Severe trauma and associated musculoskeletal injuries result in the acute release of Damage-Associated Molecular Patterns (DAMPs) in plasma, many of which are made of nucleic acids. DAMPs then bind leukocytes and trigger NETosis (Neutrophil Extracellular Traps), the release of nuclear material coated with proteolytic enzymes, which ultimately promotes remote lung injury and acute respiratory distress syndrome (ARDS).

Considering that many DAMPs and all NETs are made of nucleic acids, we hypothesize that dornase alfa, a commercially available recombinant desoxyribonuclease (DNAse) could reduce DAMPs and NETs-induced lung injury in severe trauma patients under mechanical ventilation in the intensive care unit (ICU).

The primary objective is to demonstrate a reduction in the incidence of moderate to severe ARDS in severe trauma patients during the first seven ICU days from 45% to 30% by providing aerosolized dornase alfa once during the first two consecutive ICU days and compared to equivalent provision of placebo (NaCl 0,9%).

The secondary objectives are to demonstrate, by using aerosolized dornase alfa compared to placebo:

* an improvement in static lung compliance
* a reduction in mechanical ventilation duration / an increase in ventilation-free ICU days
* a reduction in the length of ICU stay
* a reduction in the hospital length of stay
* a reduction in multi-organ failure
* a reduction in ventilator-associated pneumonia (VAP)
* a reduction in mortality at day 28

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18) patient of either sex affiliated to the National Health Service

  * Severe trauma patient (either blunt or penetrating), Injury Severity Score > 15
  * Under mechanical ventilation for an expected duration > 48h
  * Admitted in the ICU
  * Signed informed consent from the patient's relative
  * Patient equipped with an indwelling arterial catheter

Exclusion Criteria:

* Pregnancy or breast feeding

  * Opposition from the patient or his/her relatives
  * Protected major (Guardianship)
  * Contraindication to the use of dornase alfa
  * Known intolerance to dornase alfa

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-03-04 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the incidence of moderate to severe ARDS (PaO2/FiO2 < 200, according to the Berlin definition [ARDS definition task force et al. JAMA 2015; 307(23): 2526-2533]) in severe trauma patients (Injury Severity Score > 15). | Day 0 to Day 7

SECONDARY OUTCOMES:
Static lung compliance [mL/cmH2O] | Day 0 to Day 7
Duration of mechanical ventilation [hours] | Day 0 to Day 7
Length of ICU stay [hours] | Day 0 to Day 7
Length of stay in the hospital [days] | Day 0 to Day 7
Incidence of multi-organ failure | Day 0 to Day 7
  according SOFA (Sepsis-related Organ Failure Assessment) to quantify organ dysfunction
Incidence of Ventilator-Associated Pneumonia (VAP) | Day 0 to Day 7
Mortality on day 28 | Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Strasbourg, france, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pottecher J, Noll E, Borel M, Audibert G, Gette S, Meyer C, Gaertner E, Legros V, Carapito R, Uring-Lambert B, Sauleau E, Land WG, Bahram S, Meyer A, Geny B, Diemunsch P. Protocol for TRAUMADORNASE: a prospective, randomized, multicentre, double-blinded, placebo-controlled clinical trial of aerosolized dornase alfa to reduce the incidence of moderate-to-severe hypoxaemia in ventilated trauma patients. Trials. 2020 Mar 18;21(1):274. doi: 10.1186/s13063-020-4141-6. PMID 32183886